CLINICAL TRIAL: NCT06072729
Title: "Comparison of Magnesium Sulphate Versus Cold Compression on Patients With I.V Cannula Induce Phlebitis Admitted in Lahore General Hospital Lahore a Randomized Control Trial
Brief Title: Comparison of Magnesium Sulphate Versus Cold Compress in IV Cannula Induces Phlebitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Nadia Manzoor, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cold compression 1507
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Patient With IV Cannula Induce Phlebitis
Keywords: comparison, Magnesium Sulphate, Cold Compress, Phlebitis
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesuuim Sulphate (Experimental): After the initial assessment, the cannula will be removed from the site (if present) the cannulation site will be cleaned with normal saline. A mixture of 100mg magnesium sulfate and glycerin will be applied to a gauze pad (2" × 2"). This gauze pad placed on the site of phlebitis induced by peripheral intravenous catheter (PIVC). This will be done three times a day for three consecutive days
  Interventions: Other: comparison of magnesium sulphate versus cold compression
- Cold compression (Experimental): After the initial assessment, the cannula will be removed from the site (if present) and the area will be cleaned with normal saline. A gauze pad (2" × 2") soaked in cold water with a temperature below 15 °C will be applied to the phlebitis site for 20 minutes. This will be done three times a day for three consecutive days. The cold water will be stored in the refrigerator in the respective wards one day prior to the dressing. It will be taken from the refrigerator just before the dressing and applied within one minute. After 20 minutes of application, the gauze pad for cold compress will be removed from the phlebitis site. From 1st to 3rd Day daily assessment done through VIP scale, will be conducted in both Group A (magnesium sulphate group) and Group B (cold compression group)
  Interventions: Other: comparison of magnesium sulphate versus cold compression

INTERVENTIONS:
Other: comparison of magnesium sulphate versus cold compression — This study will involve a total of 70 participants who will be divided into two groups. One group will receive magnesium sulphate, while the other group will receive cold compression. The severity of phlebitis will be assessed in both groups using a visual phlebitis (VIP) rating scale.
  Other Names: cold comprssion

SUMMARY:
The use of intravenous (IV) devices is an integral part of patient care in hospitals, clinics, maternity home etc. approximately 80% of hospitalized patients receive I.V therapies. Phlebitis is a complication that is frequently associated with intravenous therapy. Phlebitis is the inflammation of a vein. It most commonly occurs in superficial veins. It is characterized by local pain, tenderness, swelling, induration, and erythema of the venous tract, and a palpable cord-like vein on the infusion site. The most common causes of phlebitis may be mechanical, chemical, and bacterial. Phlebitis may lead to life-threatening complications such as pain, Cellulitis, gangrene and it leads to amputation of the limb. The possibility of clot formation in the veins can lead to serious complications such as deep vein pulmonary embolism, which can cause sudden death. Other complications include septic shock, thrombophlebitis requiring supportive treatment, metastatic infection, the formation of liver abscesses, and endocarditis due to septic emboli. Patients with chronic diseases like diabetes, coronary heart disease, renal failure, hepatic encephalopathy, neurological conditions, and those who are bedridden for extended periods, as well as newborns, face difficulties in maintaining intravenous (IV) cannulas. As a result, needs to maintain central lines for fluids and medication, which is another source of infection. These complications can lead to prolonged hospital stays, increased medical costs, reduced patient satisfaction, and a lower quality of life for the affected individuals. Here the question arises for nurses to check the effectiveness of magnesium sulphate versus cold compress. To find the answer to this question this study will be conducted with the objective of comparing magnesium sulfate versus cold compression on patients with a peripheral intravenous cannula (PIVC) induced phlebitis, hospital-based comparative study and the simple random sampling technique will be used to collect a sample of sixty participants and will be equally distributed into two groups. The study will be conducted in Lahore general hospital Lahore Punjab Pakistan.

DETAILED DESCRIPTION:
Materials & Methods/Subjects & Methods:

Study Design:

• This study will be a Randomized Control Trial.

Setting:

This study will be carried out at the Institute of Nursing University of Health Sciences, Lahore in the collaboration with Lahore General Hospitals Lahore, Pakistan which is one of the major teaching hospitals and sample will be collected from Medical units, surgical units.

Duration:

The anticipated duration of this study will be 12 months.

Sample Size:

The sample size for each group is 35 calculated by using the following formula with estimated 80% power of the study, 95% confidence interval, and assuming that of phlebitis in group1: 96.70% and group 2 is 76.7% (Hongmei et al., 2020) (Sample size is calculated through the WHO online calculator)

Sampling Technique:

A total of 70 patients will be selected by simple random sampling. The patients will be randomized into two groups by lottery method. Group 1 (magnesium sulfate application) and Group 2 (cold compression) will be given. In this method, 70 cards having the same appearance will be used, 35 of them with letter 1 for group 1 and other letter 2 for group 2. Each participant should take one card from this box. Therefore random allocation of subjects will be determined (Dahal et al., 2020).

ELIGIBILITY:
Inclusion Criteria:

The patient admitted for 72 hours or more than 72 hours.

* Patient with intravenous therapy.
* Patients with signs of phlebitis 2-4 score on the VIP scale.
* Age group of 18-50 years and able to report pain.

Exclusion Criteria:

* Patient with superficial thrombophlebitis and having skin disorder.
* Patient having associated muscular disorders like DVT, varicose veins,s, etc.
* Patient with disturbed coagulation profile.
* I.V Drug abusers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of phlebitis score | 3 days 3 time a day
  magnesium sulphate and cold compression reduce the phlebitis score

IPD SHARING:
Plan to Share IPD: No